CLINICAL TRIAL: NCT02339415
Title: Targeted Anticoagulation Therapy to Reduce Inflammation and Cellular Activation in Long-term HIV Disease
Acronym: TACTICAL-HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Jason Baker, Protocol Chair, Hennepin Healthcare Research Institute
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCC-008
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Inflammation; Coagulation; HIV Infection
MeSH Terms: conditions — Inflammation; Thrombosis; HIV Infections | interventions — edoxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): Edoxaban 30mg daily
  Interventions: Drug: Edoxaban 30mg daily
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Edoxaban 30mg daily
  Arms: Treatment
Drug: Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of pharmacologic FXa inhibition (via edoxaban 30 mg daily) on inflammation, as reflected in plasma Interleukin-6 levels.

DETAILED DESCRIPTION:
We hypothesize that increased generation of activated factor X (FXa) contributes to a systemic elevation in pro-inflammatory cytokine levels (e.g. IL-6) among HIV positive patients. This occurs, in part, via FXa activation of protease activated receptor 2 (PAR-2) on monocytes and tissue macrophages, which perpetuates innate inflammation. We will test our hypothesis with an oral antagonist to FXa (edoxaban), and quantify the immunologic effects of PAR-2 inhibition on systemic inflammation and monocyte activation.

The potential benefits of pharmacologic inhibition of FXa will be studied among HIV positive participants receiving ART with suppressed HIV viral load and a D-dimer >100 ng/mL. The study design is a cross-over placebo controlled randomized trial of edoxaban 30mg daily versus matched placebo (n=40 total participants). After screening and baseline visits, participants will be randomized to the sequence of drug administration (i.e., edoxaban vs. placebo). After randomization, participants will start study medication #1 and follow-up for visits at months 1, 2, 3 and 4. They will then stop study medication for 3 months, return for visits at months 7 and 8 (analogous to screening and baseline, respectively), then start study medication #2 and follow-up for visits at months 9, 10, 11, and 12.

The treatment effect (i.e., changes from pre-treatment levels) over 4 months will be assessed in measures of inflammation, immune activation, and coagulation. For comparisons with placebo, each participant will then serve as his or her own control in this cross-over design.

ELIGIBILITY:
Inclusion Criteria

* HIV infection (verified by previous positive antibody or detectable HIV RNA level)
* Age ≥18 years
* Receiving continuous ART for ≥2 years (regimen changes >3 months prior to enrollment are acceptable)
* HIV RNA level ≤200 copies/mL for ≥1 year (1 measure ≥200 allowed if also <500 and preceded and followed by one or more values ≤200 copies/mL)
* D-dimer level ≥100 mg/L (or ng/mL) at screening (or within the prior month)
* Estimated creatinine clearance ≥50 mL/min
* Body weight ≥60kg
* Do not anticipate starting (or stopping) statin or aspirin therapy during the study
* For women of child bearing potential, agrees to use a reliable form of birth control

Exclusion Criteria

* Pregnancy or breast feeding
* A contra-indication to taking edoxaban
* A clinical indication for anticoagulation therapy (e.g., atrial fibrillation or Deep Vein Thrombosis/PE)
* Treatment with anti-platelet, anti-coagulation, or immune-modulatory drugs currently or within the past 6 months; prior self-limited treatment with aspirin (i.e., not daily use) is not itself an exclusion.
* Grade ≥1 hematology lab abnormality for INR (>1.1 x ULN), hemoglobin (<10.0 g/L), platelets (<100,000 cells/μL), and WBC (2,500 cells/mm3)
* Grade ≥2 lab abnormality for chemistries (BMP) or liver panel
* Alcohol or illicit drug abuse/dependency within the prior year
* History of prior myocardial infarction or unstable atherosclerotic disease
* History of prior stroke or transient ischemic attack (TIA)
* History of active gastrointestinal ulcer or bleeding disorder within the prior year
* Intent to have surgery during the study period (12 months)
* Hepatitis C treatments (e.g., interferon, ribavirin, protease inhibitors) within the past 6 months
* Cirrhosis or hepatic impairment (e.g., Child-Pugh class B or C).
* Seizure disorder
* Previous/current CNS space occupying lesion (e.g., Toxoplasmosis, mTB) with persistent abnormalities on CNS imaging after completion of treatment.
* Surgical or invasive procedure anticipated during study period.
* Invasive cancer in the prior year or receiving cancer treatment (not including carcinoma-in-situ or basal cell cancer of the skin)
* Rheumatologic or inflammatory disease, systemic in nature (e.g., systemic lupus erythematosus, rheumatoid arthritis, vasculitis, sarcoidosis, Crohn's disease)
* Assessment by the clinical investigator that enrollment into the study could entail excess risk to the participant, beyond what is intended or expected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Baker, M.D., Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First Then Edoxaban: Participants receive placebo during first period, then Edoxaban (30mg daily) in second period after washout.
- Edoxaban First Then Placebo: Participants receive Edoxaban (30mg daily) in first period, then placebo during second period after washout.
Period: First Period
Arm/Group | Placebo First Then Edoxaban | Edoxaban First Then Placebo
Started | 22 | 22
Received at Least One Dose | 21 | 20
Completed | 20 | 20
Not Completed | 2 | 2
Period: Washout
Arm/Group | Placebo First Then Edoxaban | Edoxaban First Then Placebo
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Second Period
Arm/Group | Placebo First Then Edoxaban | Edoxaban First Then Placebo
Started | 20 | 20
Completed | 19 | 18
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First Then Edoxaban | Edoxaban First Then Placebo | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (8) | 47 (10) | 49 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 18 | 22 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black | 8 | 2 | 10
  Hispanic or Latino | 1 | 1 | 2
  White (Non-Hispanic) | 13 | 18 | 31
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 122.4 (17.3) | 126.1 (13.0) | 124.3 (15.3)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 81.4 (11.0) | 78.9 (10.4) | 80.1 (10.6)
Interleukin-6 (IL-6) [Median (Inter-Quartile Range); unit: pg/mL] | 0.695 [0.520 to 1.080] | 0.465 [0.380 to 0.980] | 0.575 [0.395 to 1.020]
D-dimer [Median (Inter-Quartile Range); unit: μg/mL] | 0.18 [0.11 to 0.24] | 0.18 [0.13 to 0.34] | 0.18 [0.12 to 0.31]

OUTCOME MEASURES:

1. Primary Outcome: Change in Interleukin 6 (IL-6) Plasma Levels From Baseline to 4 Months.
Description: Difference between treatment and control ln-transformed IL-6 plasma levels in change from pre-treatment to on-treatment values
Time Frame: Through study completion, an average of 4 months on each treatment.
Population: 44 participants were randomized to each arm, of those, 41 went on to receive placebo and have follow up data, 40 received study drug (Edoxaban) and had follow up data.
Measure: Mean (Standard Deviation); unit: ln-pg/mL
Groups:
- Placebo: Matched placebo
- Edoxaban: 30mg of Edoxaban
Arm/Group | Placebo | Edoxaban
Number analyzed (Participants) | 41 | 40
ln-pg/mL | -0.02 (0.39) | 0.09 (0.29)
Statistical Analysis 1: Comparison: Placebo vs Edoxaban; Test type: Superiority; p = 0.26, Mixed Models Analysis; included predictors: treatment, assigned treatment sequence and pre-treatment biomarker level; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.06 to 0.21], Standard Error of Mean 0.07 — because biomarkers were analyzed on natural log scale, the estimated parameter is the log-transformed mean percent difference in treatment effect on Edoxaban vs. Placebo

2. Secondary Outcome: Change in D-Dimer Levels From Baseline to 4 Months
Description: Difference between treatment and control ln-transformed D-Dimer levels in change from pre-treatment to on-treatment values
Time Frame: Through study completion, an average of 4 months on each treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ln-μg/mL
Arm/Group | Placebo | Edoxaban
Number analyzed (Participants) | 41 | 40
ln-μg/mL | -0.13 (0.77) | -0.66 (1.01)
Statistical Analysis 1: Comparison: Placebo vs Edoxaban; Test type: Superiority; p = 0.002, Mixed Models Analysis; included predictors: treatment, assigned treatment sequence and pre-treatment biomarker level; Mean Difference (Net) = -0.54, 95% CI 2-sided [-0.88 to -0.20], Standard Error of Mean 0.17 — [estimate comment as in outcome 1, analysis 1]

3. Other Pre Specified Outcome: Safety (Bleeding Events)
Description: Number of bleeding events on Edoxaban or Placebo.
Time Frame: 4 months while on Edoxaban or Placebo
Measure: Number; unit: event
Groups:
- Receiving Placebo: Administered matched placebo
- Receiving Edoxaban: Administered 30mg of Edoxaban
Arm/Group | Receiving Placebo | Receiving Edoxaban
Number analyzed (Participants) | 44 | 44
event
  Epistaxis | 2 | 8
  Bruising | 5 | 7
  Bleeding gums | 3 | 10
  Bloody stool | 3 | 4
  Hematuria | 0 | 1
  Laceration | 2 | 5

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Placebo | Edoxaban
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/44 | 1/44
Other Adverse Events (participants affected / at risk) | 21/44 | 21/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=44) | Edoxaban (N=44)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=44) | Edoxaban (N=44)
Viral Gastroenteritis (Gastrointestinal disorders) | 0 | 1 (1)
Vomiting and Diarrhea (Gastrointestinal disorders) | 0 (0) | 1
cut head, slipped on ice (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Iron Deficiency Anemia, unspecified iron deficiency anemia type (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ruptured L5 disc (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Grade 3 AST due to HCV seroconversion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Grade 4 ALT due to HCV seroconversion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Bleeding from a minor dog bite (puppy) with unusual bruising (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hit by softball, bleeding from eye laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration secondary to coffee pot (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration secondary to meat slicer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
hematuria (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
exhaustion (General disorders) | 0 (0) | 1 (1)
Acute macular neuroretinopathy (Eye disorders) | 0 (0) | 1 (1)
Laceration secondary to syncope (General disorders) | 1 (1) | 0 (0)
Motor vehicle accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lightheadedness (General disorders) | 3 (3) | 0 (0)
Osteoporosis diagnosis via DEXA on routine clinical screening (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Severe back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bleeding of minor cuts/slow healing (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
bleeding gums (Blood and lymphatic system disorders) | 3 (3) | 7 (10)
Blood in stool (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Epistaxis (Blood and lymphatic system disorders) | 2 (2) | 5 (8)
Bruising (Blood and lymphatic system disorders) | 5 (5) | 7 (7)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 0 (0)
Dizziness (General disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT02339415/Prot_SAP_ICF_000.pdf